CLINICAL TRIAL: NCT00101361
Title: CSP #535 - Anabolic Steroid Therapy on Pressure Ulcer Healing in Persons With Spinal Cord Injury
Brief Title: Oxandrolone to Heal Pressure Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility analysis showed low probability of detecting a significant difference
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 535
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Pressure Ulcer
Keywords: dermatologic; skin; clinical trial; androgen/anabolic
MeSH Terms: conditions — Pressure Ulcer | interventions — Oxandrolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oxandrolone
  Interventions: Drug: Oxandrolone
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxandrolone — Patients will receive oxandrolone (10mg BID) until full healing occurs or for 24 weeks, which ever comes first.
  Arms: 1
Drug: Placebo — Patients will receive an identically appearing placebo capsule until full healing occurs or for 24 weeks, which ever comes first.
  Arms: 2

SUMMARY:
This study is designed to determine whether the use of oxandrolone, an anabolic steroid, can heal pressure ulcers in persons with spinal cord injury (SCI). In a Feasibility Study, three VA SCI Units will screen and randomize patients into treatment with oxandrolone or with placebo. Eleven other sites will screen patients to determine eligibility but will not treat patients with the agent. Following the Feasibility Study, all sites will participate in a blinded, randomized treatment study. A total of 400 patients will be enrolled over a four-year period. Any patient in a participating unit who has chronic SCI and a difficult-to-heal pelvic ulcer will be eligible for the study if other entry criteria are met. All enrolled patients will be followed for a period of 24 weeks to determine whether their target pressure ulcers heal. Those who are healed will be followed for an additional four weeks to determine whether the ulcer remains healed.

DETAILED DESCRIPTION:
The primary objective is to determine whether SCI inpatients with a chronic Stage III or IV pressure ulcer of the pelvic region who are randomized to receive 24 weeks of optimized clinical care and an oral anabolic steroid agent (oxandrolone) will have a greater percent of healed pressure ulcers than those who receive placebo and the same optimized clinical care. The major secondary objective is to determine whether the healed pressure ulcer will remain healed for at least 8 weeks.

Subjects are registered into a 4 week screening phase to be followed with weekly photos of the ulcer and if healed less than 30% (from the day 1 photo to the day 28 photo) with standard clinical care, they are introduced to the treatment phase (randomized) and followed for another 24 weeks on either oxandrolone or placebo. Wounds that heal (remain closed for at least 96 hours) are then subject to 2 four week follow up visits.

Criteria for entering the screening phase are simple: either gender, age 18 years or older, inpatient with SCI or equivalent spinal cord damage and at least 1 Stage III or IV (indicating a severe wound, <260cm2) pressure ulcer of the pelvic region.

September 2006 - year one report submitted and approved by Central Office. Plan to add up to 3 more sites in the next year.

January 2007 - site #16 (San Antonio) is approved by Veterans Affairs Cooperative Studies Program Central Office to be invited.

ELIGIBILITY:
Inclusion Criteria:

SCREENING PHASE:

1. Male or female inpatient with SCI or equivalent spinal cord damage.
2. At least one Stage III or IV (including a severe wound, <260cm2) pressure ulcer of the pelvic region.

TREATMENT PHASE:

1. documentation (through screening phase) of difficult to heal (defined as <30% area reduction) or worsening status of the pressure ulcer for at least 28 days as inpatient (screening phase)

Exclusion Criteria:

SCREENING PHASE:

1. Persons who are candidates for and elect to have reconstructive flap surgery of the TPU;
2. Persons with known osteomyelitis who have not been, or refuse to be, adequately treated with appropriate antibiotic treatment for at least 6 weeks and/or appropriate surgical procedures, as determined by the patients' physician, as well as patients who have not had resolution of osteomyelitis after 3 months of antibiotic and/or surgical care.
3. Psychopathology (documentation in the medical record or history of self-abusive behavior specific to pressure ulcer healing which may or may not include major or minor psychiatric illness) that may conflict with study objectives;
4. Previously diagnosed active malignant disease;
5. Suspicion of skin cancer at the pressure ulcer site (a biopsy-negative patient is not excluded, nor is a biopsy-positive patient excluded after a curative excision of the lesion);
6. Radiation therapy in the pressure ulcer field at anytime during the patient's lifetime;
7. Life expectancy less than 12 months;
8. Nephrosis, hemodialysis or chronic ambulatory peritoneal dialysis therapy;
9. AIDS patients at immunological risk of infectious complications defined as any of the following: (1) CD4 count <100 cells/ L or (2) CD4 count 100 to 200 cells/ L and WBC < 4,000 cells/ L or (3) a confirmed viral load within the past 6 months;
10. Administration of oxandrolone or another anabolic agent (not including testosterone replacement therapy) within the past 6 months;
11. A known hypersensitivity to anabolic steroid medications (specifically oxandrolone);
12. Coronary athersclerosis with unstable angina pectoris or a history within the past 3 months of an acute myocardial event or decompensated congestive heart failure.
13. Inability or unwillingness of the subject or surrogate to provide informed consent.

TREATMENT PHASE:

1. TPU >200 cm2 surface area of the pelvic region
2. Pressure ulcers with a clinical impression that are not expected to heal, such as those with: osteomyelitis (defined as persons with known osteomyelitis who have not been, or refuse to be, adequately treated with appropriate antibiotic treatment for at least 6 weeks and/or appropriate surgical procedures, as determined by the patients' physician, as well as patients who have not had resolution of osteomyelitis after 3 months of antibiotic and/or surgical care), sinus tracts suggestive of active osteomyelitis, communication to the synovial space, or other conditions;
3. Patient had flap surgery of the TPU during the Screening Phase;
4. Multiple full-thickness pressure ulcers that have a body surface area totaling >500cm2;
5. Clinical and/or laboratory evidence suggestive of prostate cancer;
6. Elevated liver function tests (AST >112 IU/L or bilirubin >3mg/dl);
7. Diabetes mellitus with less than optimal glycemic control (HbA1c >8.0%);
8. Received moderate (equivalent to prednisone 40 to 60 mg/d) or high dose (equivalent to prednisone >60 mg/d) systemic corticosteroids for at least 4 weeks, immunosuppressive agents, anti-cancer agents, or any radiation therapy within 30 days prior to randomization or are likely to receive one of these therapies during study participation;
9. Initiating or continuing therapy with appetite stimulants (e.g., Megase);
10. Current pharmacological therapy for hepatitis B or C infection;
11. Pregnancy or lactating female;
12. Females of child-bearing potential who are unwilling to agree to abstinence from sexual intercourse or the use of two reliable forms of contraception during the study; males unwilling to agree to abstinence from sexual intercourse or use of a condom during the study;
13. Expected use of oral anticoagulants (e.g. warfarin sodium) during the treatment phase;
14. Hypercalcemia;
15. Coronary athersclerosis with unstable angina pectoris or a history within the past 3 months of an acute myocardial event or decompensated congestive heart failure;
16. Participation in another active treatment clinical trial;
17. Inability or unwillingness of the subject or surrogate to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Study Chair — VA Medical Center, Bronx
Locations (16):
- United States (15):
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, Miami, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA Medical Center, Bronx, The Bronx, New York
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Derived] Bauman WA, Spungen AM, Collins JF, Raisch DW, Ho C, Deitrick GA, Nemchausky BA, Goetz LL, Park JS, Schwartz M, Merritt JL, Jayawardena V, Sandford P, Sabharwal S, Holmes SA, Nasar F, Sasaki R, Punj V, Zachow KF, Chua WC, Thomas MD, Trincher RC. The effect of oxandrolone on the healing of chronic pressure ulcers in persons with spinal cord injury: a randomized trial. Ann Intern Med. 2013 May 21;158(10):718-26. doi: 10.7326/0003-4819-158-10-201305210-00006. PMID 23689765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrollment started 08/01/2005 and ended 10/10/2008 at 15 VA Medical Centers. Subjects were randomized only after a four week screening phase.
Pre-assignment Details: Potential participants were screened for four weeks to determine eligibility based on documentation of a difficult-to-heal or worsening status of the pressure ulcer as an inpatient.
Groups:
- 1 Oxandrolone: oxandrolone - two 5mg capsules twice daily
- 2 Placebo: placebo - two capsules twice daily
Period: Overall Study
Arm/Group | 1 Oxandrolone | 2 Placebo
Started | 108 | 104
Completed | 108 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: overall baseline participants were determined by number of participants that were eligible after screening based on a pressure ulcer that is defined as hard-to-heal or worsening at randomization.
Groups:
- Oxandrolone: Oxandrolone
- Placebo: placebo
- Total: Total of all reporting groups
Arm/Group | Oxandrolone | Placebo | Total
Number analyzed (Participants) | 108 | 104 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 83 | 165
  >=65 years | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.4) | 57.3 (11.6) | 57.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 106 | 104 | 210
Region of Enrollment [Number; unit: participants]
  United States | 107 | 103 | 210
  Puerto Rico | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: A Healed Pressure Ulcer
Description: Patients remained in treatment until full healing of the target pressure ulcer (defined as re-epithelialization to a cicatrix with a dry surface and zero open area for a minimum of 96 hours) or 24 weeks, whichever occured first.
Time Frame: healing was measured from randomization to full healing or 24 weeks, whichever occured first.
Measure: Number; unit: participants
Arm/Group | 1 Oxandrolone | 2 Placebo
Number analyzed (Participants) | 108 | 104
participants | 26 | 31
Statistical Analysis 1: Comparison: 1 Oxandrolone vs 2 Placebo; For spinal cord injury patients with a Stage III or IV pressure ulcer of the pelvic region who receive 24 weeks or less of optimized clinical care (i.e., guideline-driven care with nutritional support) compared with optimized clinical care and an oral anabolic steroid agent (oxandrolone) there will be no difference in the percent of healed pressure ulcers; Test type: Non-Inferiority or Equivalence — the required sample size of 400 participants provided 85% power to detect an increase in healing from 25% in the placebo group to 40% in the oxandrolone group, as assuming a 0.05 (2-sided) type I error, 13% rate of loss to follow up, and a test of proportions by using an arcsine transformation; p < 0.05, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-17.5 to 6.8]

ADVERSE EVENTS:
Time Frame: years, 5 months
Description: Adverse events were reported for each event not each subject, therefore participants could have one or more events. The total events as reported is expected to surpass the total participants. The total participants with at least one adverse event (AE) is 95 oxandrolone and 85 placebo.
Arm/Group | 1 Oxandrolone | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 9/108 | 16/104
Other Adverse Events (participants affected / at risk) | 95/108 | 85/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1 Oxandrolone (N=108) | 2 Placebo (N=104)
oral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
small bowel obstruction, renal failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
elective bladder stone removal (Surgical and medical procedures) | 1 (1) | 0 (0)
myocutaneous flap surgery (Surgical and medical procedures) | 5 (5) | 9 (9)
death (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
death (Respiratory, thoracic and mediastinal disorders) | 3/104 (3) | 3 (3)
death (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Oxandrolone (N=108) | 2 Placebo (N=104)
anemia (Blood and lymphatic system disorders) | 17 (17) | 4 (4)
constipation or diarrhea (Gastrointestinal disorders) | 8 (8) | 10 (10)
elevated liver enzyme levels (Investigations) | 35 (35) | 3 (3)
fever (Injury, poisoning and procedural complications) | 17 (17) | 10 (10)
infection (Infections and infestations) | 13 (13) | 9 (9) — cellulitis, sepsis, clostridial
nausea / vomitting (Gastrointestinal disorders) | 10 (10) | 10 (10)
non-Target Pressure Ulcer (TPU) skin ulcer (Skin and subcutaneous tissue disorders) | 13 (13) | 8 (8)
osteomylitis (Infections and infestations) | 5 (5) | 6 (6)
pneumonia (Infections and infestations) | 14 (14) | 6 (6)
skin rash / complication (Skin and subcutaneous tissue disorders) | 15 (15) | 10 (10)
urinary tract infection (Infections and infestations) | 37 (37) | 28 (28)

LIMITATIONS AND CAVEATS:
Selection of severe wounds may have reduced treatment response. The study was terminated after a futility analysis showed a low probability of detecting a significant difference between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes